CLINICAL TRIAL: NCT01579760
Title: Treatment of Radiation Retinopathy With Intravitreal Aflibercept Injection 2.0mg
Brief Title: Intravitreal Aflibercept Injection for Radiation Retinopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aflibercept2012
Record Dates: First submitted 2012-04-10; First posted 2012-04-18 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Radiation Retinopathy; Macular Edema
Keywords: radiation; retinopathy; macular edema; anti-VEGF; VEGF-Trap; aflibercept
MeSH Terms: conditions — Macular Edema; Retinal Diseases | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aflibercept every 2 months (Experimental)
  Interventions: Drug: Aflibercept every 2 months
- aflibercept monthly (Experimental)
  Interventions: Drug: Aflibercept monthly

INTERVENTIONS:
Drug: Aflibercept every 2 months — 2.0 mg aflibercept intravitreal injections once per month for the first 3 months (M0, M1, M2), then every 2 months (M4, M6, M8, M10)
  Other Names: EYLEA; VEGF Trap-Eye
  Arms: aflibercept every 2 months
Drug: Aflibercept monthly — 2.0mg aflibercept intravitreal injections every month (M0-11)
  Other Names: EYLEA; VEGF Trap-Eye
  Arms: aflibercept monthly

SUMMARY:
The purpose of this study is to assess the safety of intravitreal aflibercept injection - in the treatment of macular edema associated with retinopathy secondary to previous radiation therapy.

DETAILED DESCRIPTION:
Radiation retinopathy can cause decreased vision in patients who have received either external beam radiation or local plaque therapy to the eye. An early manifestation of radiation retinopathy is macular edema, which represents fluid within the retina that affects central vision. There is currently no approved treatment for this disease, although there have been anecdotal reports of benefit with laser photocoagulation, intravitreal anti-VEGF agents, or intravitreal steroid use. This is a phase 1 study to evaluate aflibercept for the treatment of macular edema associated with retinopathy secondary to previous radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Retinopathy associated with previous I-125 brachytherapy for uveal melanoma (85 Gy over 96 hours) at least 6 months prior to enrollment
* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Center involved macular edema > 300µm in thickness on SD-OCT
* Best corrected visual acuity of 20/40- 20/400
* Birth control therapy for females of child-bearing age

Exclusion Criteria:

* Pre-existing retinopathy due to other disorders
* Vision decrease is considered to be due to ischemic radiation retinopathy without macular edema or optic neuropathy
* Presence of metastasis
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Prior enrollment in any study with intravitreal aflibercept injection
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Uncontrolled glaucoma in the study eye (defined as IOP ≥ 30 mmHg despite treatment with anti-glaucoma medication)
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 4 months of study enrollment.
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Any concurrent intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could either require medical or surgical intervention during the study period to prevent or treat visual loss that might result from that condition, or if allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of BCVA over the 6-month study period
* Presence of significant subfoveal fibrosis or atrophy
* Intraocular surgery (including cataract surgery) in the study eye within 2 months of enrollment
* Active intraocular inflammation (grade trace or above) in the study eye
* History of allergy to fluorescein, ICG or iodine, not amenable to treatment
* Prior/Concomitant Treatment:
* Panretinal photocoagulation treatment
* Previous intraocular steroids or PDT within 3 months
* Previous participation in any studies of investigational drugs within 30 days preceding Day 0 (excluding vitamins and minerals)
* Previous treatment with intravitreally (in either eye) or intravenously administered Avastin (bevacizumab) within 60 days or concomitant use in either eye outside the scope of this study
* Previous use of Eylea, Macugen or Lucentis in study eye within 60 days or concomitant use in either eye outside the scope of this study
* Prior submacular or vitreous surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-11; Primary Completion 2019-01 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 12 months
Severity of adverse events | 12 months

SECONDARY OUTCOMES:
Mean change in best corrected visual acuity from baseline | 12 months
Mean change in central foveal thickness by optical coherence tomography (OCT) from baseline | 12 months
Mean visual acuity | 12 months
Mean central foveal thickness | 12 months
Proportion of patients gaining 3 lines of vision | 12 months
Mean change in lesion characteristics (lesion size, leakage) | 12 months
Proportion of patients with no fluid on OCT | 12 months
Mean change in macular volume | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Prabakar K Rao, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Retina Consultants of Houston, Houston, Texas

REFERENCES:
- [Background] Horgan N, Shields CL, Mashayekhi A, Teixeira LF, Materin MA, Shields JA. Early macular morphological changes following plaque radiotherapy for uveal melanoma. Retina. 2008 Feb;28(2):263-73. doi: 10.1097/IAE.0b013e31814b1b75. PMID 18301032
- [Background] Finger PT, Chin K. Anti-vascular endothelial growth factor bevacizumab (avastin) for radiation retinopathy. Arch Ophthalmol. 2007 Jun;125(6):751-6. doi: 10.1001/archopht.125.6.751. PMID 17562985
- [Background] Wen JC, McCannel TA. Treatment of radiation retinopathy following plaque brachytherapy for choroidal melanoma. Curr Opin Ophthalmol. 2009 May;20(3):200-4. doi: 10.1097/ICU.0b013e328329b62d. PMID 19349865